CLINICAL TRIAL: NCT00953641
Title: Vaginal Misoprostol for Cervical Ripening Prior to Endometrial Biopsy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Principle Investigator retired, Resident moved away
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Anita Harding, Dr., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-134
Record Dates: First submitted 2008-08-26; First posted 2009-08-06 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Menorrhagia; Endometrial Biopsy; Cervical Ripening
Keywords: Vaginal Misoprostol; Cervical ripening; Endometrial biopsy
MeSH Terms: conditions — Menorrhagia | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pre-Menopausal 1 (Active Comparator): Pre-Menopausal group, receiving Misoprostol
  Interventions: Drug: Misoprostol
- Pre-Menopausal 2 (Placebo Comparator): Patients will insert a placebo vaginal suppository 12h or more prior to the endometrial biopsy
  Interventions: Drug: Placebo
- Post-Menopausal 1 (Active Comparator): Post-Menopausal patients will insert a Misoprostol vaginal suppository 12h or more prior to the endometrial biopsy
  Interventions: Drug: Misoprostol
- Post-Menopausal 2 (Placebo Comparator): Placebo vaginal suppository prior to the endometrial biopsy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — Misoprostol 400ug, suspended in a base (Witepsol 15) as a vaginal suppository Single dose 12h or more prior to the procedure
  Other Names: Cytotec
  Arms: Post-Menopausal 1; Pre-Menopausal 1
Drug: Placebo — Witepsol 15 base, vaginal suppository, Single dose, 12h or more prior to the endometrial biopsy
  Arms: Post-Menopausal 2; Pre-Menopausal 2

SUMMARY:
The purpose of this study is to determine whether using Misoprostol vaginally before an office endometrial biopsy is performed, will make it easier, more successful and less painful to do the procedure.

The investigators' hypothesis is that vaginal Misoprostol 12 hours prior to endometrial biopsy will increase the ease of performing office endometrial biopsy by reducing the need to use a tenaculum or a cervical dilator to achieve passage of a biopsy pipelle.

DETAILED DESCRIPTION:
Endometrial biopsy is a common gynecological office procedure performed to assist in the pathological diagnosis of abnormal vaginal bleeding. The procedure can be painful and it may be difficult to obtain an endometrial sample with a hard and closed cervix. Giving Misoprostol before the procedure may soften the cervix sufficiently to allow an easier and more successful test. This medication has been tested before hysteroscopy and in some patients it has been shown to be beneficial.

104 patients need to be recruited for this study. Participants will be divided according to pre-menopausal and post-menopausal status. Each of these groups will then be divided into a treatment arm (with Misoprostol) and a placebo arm. Participants will place a vaginal suppository containing either Misoprostol 400 ug or a placebo 12h or more before their appointment for the endometrial biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with abnormal uterine bleeding
* Age over 35 years

Exclusion Criteria:

* Pregnancy
* Allergy to or contraindication to prostaglandin use
* Active genital tract infections
* Bleeding disorders

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Evaluating the ease of an endometrial biopsy by the need to use a tenaculum or a cervical dilator to achieve passage of a biopsy pipelle | 1 year

SECONDARY OUTCOMES:
Evaluating participants discomfort during the procedure, using a pain scale | 1 year
Success rate of passage of the pipelle | 1 year
Adverse effects from medications | 1 year
Complications of the procedure | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Roger Pierson, PhD, Study Chair — University of Saskatchewan, Dept. of Obstetrics and Gynecology, College of Medicine; Anita Harding, MBChB, Principal Investigator — University of Saskatchewan, Dept. of Obstetrics and Gynecology, College of Medicine; Thirza Smith, MD, FRCS, Principal Investigator — University of Saskatchewan, Dept. of Obstetrics and Gynecology; Marilyn Davidson, FRCSC, Principal Investigator — University of Saskatchewan, Dept. of Obstetrics and Gynecology
Locations (1):
- Obstetrics and Gynecologic Consultants, Saskatoon, Saskatchewan, Canada